CLINICAL TRIAL: NCT03503513
Title: The Effect of Gentamicin Intravesical Installations on Decreasing Urinary Tract Infections in Patients With Neurogenic Bladder After Spinal Cord Injury: A Clinical Trial
Brief Title: Gentamicin Bladder Instillations to Prevent Urinary Tract Infections in Patients With Spinal Cord Injury
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Denise Tate, PhD, Professor of Physical Medicine and Rehabilitation, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HUM00137086; 90IFRE0002 (Other Grant/Funding Number: NIDRR/ACL/HHS)
Record Dates: First submitted 2018-04-06; First posted 2018-04-19 (Actual); Results first posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-05

CONDITIONS: Urinary Tract Infections; Spinal Cord Injuries; Spinal Cord Diseases; Neurogenic Bladder
MeSH Terms: conditions — Urinary Tract Infections; Spinal Cord Injuries; Spinal Cord Diseases; Urinary Bladder, Neurogenic | interventions — Gentamicins

STUDY DESIGN:
Intervention Model Description: For each participant, six month pre-treatment data is compared to data collected during treatment (count of UTIs) and immediately after treatment (self-reported measures).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gentamicin sulfate (Experimental): Participants initiate Gentamicin instillations every night for a treatment period of 6 months. Instillations are stopped if they developed a UTI. After receiving treatment for this UTI, they resume the Gentamicin instillations. After baseline screening and being consented, they are instructed on how to do the instillations through a catheter, once they receive the drug and aid equipment (i.e. syringes) to do installations. Remaining drug from syringes are to be disposed after each use. Participants use their own catheters. In-dwelling catheters are not allowed.
  Interventions: Drug: Gentamicin Sulfate

INTERVENTIONS:
Drug: Gentamicin Sulfate — Gentamicin is compounded by the Michigan Medicine Research Pharmacy in a concentration of 480 milligrams of the active product to 1000 milliliters of normal saline. Pharmacy mails participants treatment drug. Once received, participants will do daily instillations of 30 milliliters of solution after catheterizing their bladder at night.
  Other Names: Gent Instillations

SUMMARY:
A non-randomized study evaluating the efficacy of intravesical gentamicin on the occurrence rate of urinary tract infections and bladder complications in patients after spinal cord injury (SCI), and to assess its effectiveness in promoting overall quality of life (QOL), community living, and participation.

DETAILED DESCRIPTION:
Intervention: Participants' number of UTIs during the six-month treatment period will be compared to the number they incurred during the six months prior to treatment. Participants complete a baseline visit which consists of medical history, informed consent, urinalysis/culture indicating no active UTIs, metabolic panel, and self-reported measures about complications, symptoms, community participation and quality of life. Similar information is collected at the end of treatment. At a 3-month follow up visit, all available data is obtained through phone interviews and/or medical chart reviews except for self-report measures. Participants begin active treatment using Gentamicin plus saline solution after they have completed all requirements. Instillations of treatment solution occur nightly after the participant's last evening catheterization. Bi-weekly calls are conducted to ensure compliance, answer questions and document adverse events. Participants will stop the trial if they develop an UTI. After receiving treatment for the UTI by their physician, they will go into a washout period of a week before resuming the trial with Gentamicin instillations.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form and agreement to complete the daily dosing log as instructed by the study coordinator.
* History of traumatic spinal cord injury (SCI) or non-traumatic spinal cord disease, (SCD) with sustained neurological dysfunction
* At least 6 months post-initial hospital discharge following SCI/SCD onset
* Neurogenic bladder
* Ability to perform daily instillation on self or with help of others and willingness to adhere to the study regiment.
* History of at least 2 documented urinary tract infection (UTI) during the previous 6 months (prior to screening)
* Have a designated physician or health care provider for routine care
* Use of clean intermittent catheterization or catheterization through a stoma (i.e. Mitrofanoff) as their primary method of bladder management

Exclusion Criteria:

* Concurrent use of systemic oral or intravesical antibiotic prophylaxis
* Documented or self-reported history of gentamicin allergy
* Female patients who are currently pregnant or attempting to become pregnant
* Patients with a history of 8th cranial nerve disorder
* Co-morbidities like cancer and chronic disease that could impact patient safety OR significantly affect the rate of UTIs and/or quality of life (QOL) substantially
* Urological co-morbidities like bladder cancer and history of kidney disease.
* Current UTI at screening (assessed via urine analysis and culture and symptoms)
* Concurrent enrollment in a similar clinical trial
* Concurrent use of contraindicated diuretics (ethacrynic acid, furosemide)
* Current use of other contraindicated or disallowed concomitant medications or receiving treatments that may influence the results from this study.
* Known allergy to aminoglycoside antibiotics; Otological symptoms at baseline (i.e. tinnitus. severe dizziness/vertigo)
* At the discretion of study team, individuals who are unable or unlikely to comply with procedures and/or for whom study participation is not recommended (e.g. unable to arrange transportation, cognitive and/or behavioral challenges that preclude meaningful participation, poor health, etc.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise G Tate, PhD, Principal Investigator — University of Michigan; Anne Pelletier-Cameron, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 23 eligible persons who consented, only 19 started on treatment due to several reasons including changes in necessary study procedures associated with the COVID outbreak, changes in medical status due to complications and personal decisions to proceed with treatment.
Groups:
- Gentamicin Sulfate: Participants initiate Gentamicin instillations every night for a period of 6 months. Instillations are stopped if they developed a UTI. After receiving treatment for the UTI and a one week washout period, they can resume their Gentamicin instillations. After screening, being consented and completing baseline interview, participants are instructed on how to do the instillations through a catheter, once they receive the drug and aid equipment (i.e. syringes) to do installations. Remaining drug in the syringe is to be disposed after each use. Participants use their own catheters. In-dwelling catheters are not allowed.
  Gentamicin Sulfate: Gentamicin is compounded by the Michigan Medicine Research Pharmacy in a concentration of 480 milligrams of the active product to 1000 milliliters of normal saline. Participants will do daily instillations of 30 milliliters of solution
Period: Overall Study
Arm/Group | Gentamicin Sulfate
Started | 23 (consents)
Began Treatment | 19
Completed More Than 4 Months of Treatment | 12
Completed | 11
Not Completed | 12
Not completed — First cohort faced a clinical hold which caused disruption in treatment; | 4
Not completed — Second cohort faced changes due to pandemic, resulting in declining participant count | 2
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Baseline data is provided for all participants who started treatment
Groups:
- Gentamicin Sulfate: Participants initiate Gentamicin instillations every night for a period of 6 months. Instillations are stopped if they developed a UTI. After receiving treatment they can continue with the Gentamicin instillations. After baseline and consented they are instructed on how to do the instillations through a catheter, once they receive the drug and aid equipment (i.e. syringes) to do installations. Remaining drug is to be disposed after each use. Participants use their own catheters. In-dwelling catheters are not allowed.
  Gentamicin Sulfate: Gentamicin will be compounded by the Michigan Medicine Research Pharmacy in a concentration of 480 milligrams of the active product to 1000 milliliters of normal saline. Participants will do daily instillations of 30 milliliters of solution
Arm/Group | Gentamicin Sulfate
Number analyzed (Participants) | 19
Age, Continuous [Mean (Full Range); unit: years] | 46 [26 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19
Type of spinal lesions [Count of Participants; unit: Participants]
  Spinal Cord Injury (SCI) | 14
  Spinal Cord Disease (SCD) | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Urinary Tract Infections (UTI) Over Time
Description: Number of reported urinary tract infections (UTI) by participants and documented in medical chart, per person across months pre and post treatment. The number of UTIs over time was determined by establishing a per person-month rate made up of the total number of UTIs pre and during treatment (numerator) for the sample divided by the total number of persons/ 6 months (11 participants over 6 months period = 66) as the denominator. The unit of measure is defined as pre and during treatment number of UTI events per person months. These appear below under outcome measure data table.
Time Frame: 6 months prior to treatment and 6 months during treatment
Population: Eleven participants with spinal cord injury or disease and neurogenic bladder with recurrent urinary track infections (2 or more) during the 6 months prior to treatment.
Measure: Number (95% Confidence Interval); unit: UTI events per person months.
Arm/Group | Gentamicin Sulfate
Number analyzed (Participants) | 11
UTI events per person months.
  6 months prior to treatment | 0.53 [0.37 to 0.74]
  6 months during treatment | 0.09 [0.03 to 0.20]
Statistical Analysis 1: Comparison: Gentamicin Sulfate; comparison between pre and during treatment rates of UTI; Test type: Superiority; p < 0.0001, differences in incidence rate ratio; An incidence rate ratio per person/month was determined by comparing the total number of UTIs in relation to time points; Risk Ratio (RR) = 0.17, 95% CI 2-sided [0.03 to 0.20]

2. Secondary Outcome: Change in Score of Neurogenic Bladder Symptom Severity (NBSS) Scale
Description: Self-reported bladder symptoms on a scale from 0 (no symptoms) to 74 (maximum symptoms). The NBSS is a patient reported 22 item scale designed to assess symptoms and bladder related consequences among persons with neurogenic bladder dysfunction. NBSS scores are calculated across three domains with higher scores being worse and reflecting more symptoms or complications. Incontinence (scored 0-29), storage and voiding (scored 0-22), and consequences (scored 0-23). An additional question of happiness (points) was not used for this outcome.
Time Frame: Baseline to 6 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Gentamicin Sulfate
Number analyzed (Participants) | 11
score on a scale
  NBSS Incontinence (0-29) | -3.8 [-7.9 to 0.3]
  NBSS Storage/Void (0-22) | -1.1 [-3.8 to 1.7]
  NBSS Consequences (0-23) | -1.9 [-4.6 to 0.8]
Statistical Analysis 1: Comparison: Gentamicin Sulfate; NBSS Domain score for incontinence pre-post comparison; small sample size did not allow for power calculation; Test type: Superiority; p < 0.06, t-test, 2 sided — a priori threshold p value of <0.05; Mean Difference (Final Values) = -3.8, 95% CI 2-sided [-7.9 to 0.3], Standard Deviation 6.13 — Baseline to end of 6 month treatment score comparisons; (higher numbers represent more symptoms or complications)
Statistical Analysis 2: Comparison: Gentamicin Sulfate; NBSS Domain score for storage and voiding; pre-post comparison. Due to small sample size (n=11) no power calculations were conducted; Test type: Superiority; p < 0.39, t-test, 2 sided — a priori threshold p<0.05; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-3.8 to 1.7], Standard Deviation 4.09 — (higher numbers represent more symptoms or complications)
Statistical Analysis 3: Comparison: Gentamicin Sulfate; Pre and post test comparisons of mean NBSS scores for the consequences domain. Power calculations were not conducted due to small sample size; Test type: Superiority; p < 0.14, t-test, 2 sided; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-4.6 to 0.8], Standard Deviation 3.99 — Higher numbers represent more symptoms or complications referred as consequences

3. Secondary Outcome: Change in Score of Neurogenic Bowel Dysfunction (NBD)
Description: Self-reported bowel symptoms on a scale from 0 (very minor) to 14+ (severe). The NBD is a 10 item validated measure that assesses frequency of defecation and methods of bowel management and complications. Thus negative numbers in "score change" represent decrease in symptom severity.
Time Frame: Baseline to 6 months
Population: 11 participants with spinal cord injury or disease (SCI/D) with neurogenic bladder and recurrent UTIs during 6 months prior to treatment. They completed the NBD survey.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Gentamicin Sulfate
Number analyzed (Participants) | 11
score on a scale | -2.1 [-6.8 to 2.6]
Statistical Analysis 1: Comparison: Gentamicin Sulfate; Test type: Superiority; p < 0.34, t-test, 2 sided; Mean Difference (Final Values) = -2.1, 95% CI 2-sided [-6.8 to 2.6], Standard Deviation 6.99

ADVERSE EVENTS:
Time Frame: AE data was gathered for 30 days after 6 months of treatment, a total of approximately 7 months.
Arm/Group | Gentamicin Sulfate
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 4/19
Other Adverse Events (participants affected / at risk) | 17/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gentamicin Sulfate (N=19)
Renal stone removal (Renal and urinary disorders) | 1 (1)
Gross hematuria (Renal and urinary disorders) | 1 (1)
Post-COVID 19 pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
bowel obstruction (Gastrointestinal disorders) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (2)
Serratia tissue infection (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gentamicin Sulfate (N=19)
Clinically significant labs (General disorders) | 2 (2)
Urinary Tract Infection (Renal and urinary disorders) | 12 (24)
bladder spasms (Renal and urinary disorders) | 3 (6)
COVID-19 (Infections and infestations) | 4 (4)
nasal discharge (Respiratory, thoracic and mediastinal disorders) | 1 (1)
urinary discharge (Renal and urinary disorders) | 1 (1)
abdominal stoma issue (Infections and infestations) | 2 (2)
bladder irritation (Renal and urinary disorders) | 1 (1)
sweating (General disorders) | 1 (1)
heel wound (Skin and subcutaneous tissue disorders) | 2 (2)
air in bladder (Renal and urinary disorders) | 1 (1)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
bleeding from catheter site (Renal and urinary disorders) | 1 (1)
muscle strain (Injury, poisoning and procedural complications) | 1 (1)
pneumonia (Infections and infestations) | 1 (1)
flu-like symptoms (Infections and infestations) | 3 (3)
bone infection (Infections and infestations) | 1 (1)
hematuria (Renal and urinary disorders) | 1 (1)
bladder stone (Renal and urinary disorders) | 1 (1)
cystolitholapaxy (Renal and urinary disorders) | 1 (1)
GI upset (Gastrointestinal disorders) | 2 (3)
loose stool (Gastrointestinal disorders) | 1 (1)
conjunctivitis (Infections and infestations) | 1 (1)
parotitis (Infections and infestations) | 1 (1)
vaginitis (Infections and infestations) | 1 (1)
inguinal pain (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-03-09): https://cdn.clinicaltrials.gov/large-docs/13/NCT03503513/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-23): https://cdn.clinicaltrials.gov/large-docs/13/NCT03503513/SAP_002.pdf